CLINICAL TRIAL: NCT03343314
Title: Effective Management of Calcific Aortic Stenosis in the Elderly
Acronym: RAC
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 15945
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Calcific Aortic Stenosis
MeSH Terms: conditions — Aortic Valve, Calcification of

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized patients due to a severe, symptomatic aortic sten: Patients who agreed to participate in the study, aged ≥75 years, with severe and symptomatic aortic stenosis, and hospitalized in one of the medical and surgical centers participating in the study

SUMMARY:
Although aortic valve replacement is recommended for any symptomatic severe calcific aortic stenosis, the therapeutic decision may be difficult. because of patient age and comorbidities.

Transcatheter Aortic Valve Implantation (TAVI) has recently extended the therapeutic indications in patients at high risk of surgery. However, the proportion of different treatments is not known in a contemporary population that can be treated according to the different resources currently available.

The scientific goal of this observational research is to evaluate intra-hospital therapeutic decision in elderly patients referred because of symptomatic severe aortic stenosis.

The one-year survival will be analyzed according to the therapeutic decision and the characteristics of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized due to symptomatic tight aortic stenosis (NYHA >= II, dyspnea, angina or syncope);
* Having given his consent to participate in the study.

Exclusion Criteria:

* Non-severe aortic stenosis;
* Asymptomatic aortic stenosis;
* Patient under the age of 75;
* Patient refusing to participate in the study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Multicenter study to prospectively include all patients who agreed to participate in the study, with severe and symptomatic aortic stenosis, and hospitalized in one of the medical-surgical centers participating in the study and offering all the therapeutic resources for the taking into account charge of patients with aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 1101 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Collate the therapeutic decision (medical treatment, TAVI [Transcatheter Aortic Valve Implantation] or surgical aortic valve replacement) comprehensively for all hospitalized patients because of a severe, symptomatic RAC. | 1 day
  The primary endpoint is the therapeutic indication retained by the medical-surgical team in charge of the patient during hospitalization: medical treatment, TAVI or surgical aortic valve replacement.

SECONDARY OUTCOMES:
1 year-survival | 1 year
  Survival at one year will be analyzed. The analysis of the relationship between therapeutic decision and survival will be studied by taking surgical aortic valve replacement as a reference class.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iung B, Vahanian A. Epidemiology of valvular heart disease in the adult. Nat Rev Cardiol. 2011 Mar;8(3):162-72. doi: 10.1038/nrcardio.2010.202. Epub 2011 Jan 25. PMID 21263455
- [Background] Iung B, Vahanian A. Degenerative calcific aortic stenosis: a natural history. Heart. 2012 Nov;98 Suppl 4:iv7-13. doi: 10.1136/heartjnl-2012-302395. PMID 23143128
- [Background] Iung B, Cachier A, Baron G, Messika-Zeitoun D, Delahaye F, Tornos P, Gohlke-Barwolf C, Boersma E, Ravaud P, Vahanian A. Decision-making in elderly patients with severe aortic stenosis: why are so many denied surgery? Eur Heart J. 2005 Dec;26(24):2714-20. doi: 10.1093/eurheartj/ehi471. Epub 2005 Sep 1. PMID 16141261
- [Background] Bach DS, Cimino N, Deeb GM. Unoperated patients with severe aortic stenosis. J Am Coll Cardiol. 2007 Nov 13;50(20):2018-9. doi: 10.1016/j.jacc.2007.08.011. Epub 2007 Oct 29. No abstract available. PMID 17996571
- [Background] Freed BH, Sugeng L, Furlong K, Mor-Avi V, Raman J, Jeevanandam V, Lang RM. Reasons for nonadherence to guidelines for aortic valve replacement in patients with severe aortic stenosis and potential solutions. Am J Cardiol. 2010 May 1;105(9):1339-42. doi: 10.1016/j.amjcard.2009.12.056. Epub 2010 Mar 11. PMID 20403489
- [Background] Kodali SK, Williams MR, Smith CR, Svensson LG, Webb JG, Makkar RR, Fontana GP, Dewey TM, Thourani VH, Pichard AD, Fischbein M, Szeto WY, Lim S, Greason KL, Teirstein PS, Malaisrie SC, Douglas PS, Hahn RT, Whisenant B, Zajarias A, Wang D, Akin JJ, Anderson WN, Leon MB; PARTNER Trial Investigators. Two-year outcomes after transcatheter or surgical aortic-valve replacement. N Engl J Med. 2012 May 3;366(18):1686-95. doi: 10.1056/NEJMoa1200384. Epub 2012 Mar 26. PMID 22443479
- [Background] Adams DH, Popma JJ, Reardon MJ, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Buchbinder M, Hermiller J Jr, Kleiman NS, Chetcuti S, Heiser J, Merhi W, Zorn G, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Conte J, Maini B, Mumtaz M, Chenoweth S, Oh JK; U.S. CoreValve Clinical Investigators. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 May 8;370(19):1790-8. doi: 10.1056/NEJMoa1400590. Epub 2014 Mar 29. PMID 24678937
- [Background] Osnabrugge RL, Mylotte D, Head SJ, Van Mieghem NM, Nkomo VT, LeReun CM, Bogers AJ, Piazza N, Kappetein AP. Aortic stenosis in the elderly: disease prevalence and number of candidates for transcatheter aortic valve replacement: a meta-analysis and modeling study. J Am Coll Cardiol. 2013 Sep 10;62(11):1002-12. doi: 10.1016/j.jacc.2013.05.015. Epub 2013 May 30. PMID 23727214
- [Background] Martinez-Selles M, Gomez Doblas JJ, Carro Hevia A, Garcia de la Villa B, Ferreira-Gonzalez I, Alonso Tello A, Andion Ogando R, Ripoll Vera T, Arribas Jimenez A, Carrillo P, Rodriguez Pascual C, Casares i Romeva M, Borras X, Cornide L, Lopez-Palop R; PEGASO Registry Group. Prospective registry of symptomatic severe aortic stenosis in octogenarians: a need for intervention. J Intern Med. 2014 Jun;275(6):608-20. doi: 10.1111/joim.12174. Epub 2014 Mar 27. PMID 24320176
- [Background] Mylotte D, Osnabrugge RLJ, Windecker S, Lefevre T, de Jaegere P, Jeger R, Wenaweser P, Maisano F, Moat N, Sondergaard L, Bosmans J, Teles RC, Martucci G, Manoharan G, Garcia E, Van Mieghem NM, Kappetein AP, Serruys PW, Lange R, Piazza N. Transcatheter aortic valve replacement in Europe: adoption trends and factors influencing device utilization. J Am Coll Cardiol. 2013 Jul 16;62(3):210-219. doi: 10.1016/j.jacc.2013.03.074. Epub 2013 May 15. PMID 23684674
- [Background] Eltchaninoff H, Prat A, Gilard M, Leguerrier A, Blanchard D, Fournial G, Iung B, Donzeau-Gouge P, Tribouilloy C, Debrux JL, Pavie A, Gueret P; FRANCE Registry Investigators. Transcatheter aortic valve implantation: early results of the FRANCE (FRench Aortic National CoreValve and Edwards) registry. Eur Heart J. 2011 Jan;32(2):191-7. doi: 10.1093/eurheartj/ehq261. Epub 2010 Sep 15. PMID 20843959
- [Background] Gilard M, Eltchaninoff H, Iung B, Donzeau-Gouge P, Chevreul K, Fajadet J, Leprince P, Leguerrier A, Lievre M, Prat A, Teiger E, Lefevre T, Himbert D, Tchetche D, Carrie D, Albat B, Cribier A, Rioufol G, Sudre A, Blanchard D, Collet F, Dos Santos P, Meneveau N, Tirouvanziam A, Caussin C, Guyon P, Boschat J, Le Breton H, Collart F, Houel R, Delpine S, Souteyrand G, Favereau X, Ohlmann P, Doisy V, Grollier G, Gommeaux A, Claudel JP, Bourlon F, Bertrand B, Van Belle E, Laskar M; FRANCE 2 Investigators. Registry of transcatheter aortic-valve implantation in high-risk patients. N Engl J Med. 2012 May 3;366(18):1705-15. doi: 10.1056/NEJMoa1114705. PMID 22551129
- [Background] Nashef SA, Roques F, Sharples LD, Nilsson J, Smith C, Goldstone AR, Lockowandt U. EuroSCORE II. Eur J Cardiothorac Surg. 2012 Apr;41(4):734-44; discussion 744-5. doi: 10.1093/ejcts/ezs043. Epub 2012 Feb 29. PMID 22378855
- [Background] Iung B, Laouenan C, Himbert D, Eltchaninoff H, Chevreul K, Donzeau-Gouge P, Fajadet J, Leprince P, Leguerrier A, Lievre M, Prat A, Teiger E, Laskar M, Vahanian A, Gilard M; FRANCE 2 Investigators. Predictive factors of early mortality after transcatheter aortic valve implantation: individual risk assessment using a simple score. Heart. 2014 Jul;100(13):1016-23. doi: 10.1136/heartjnl-2013-305314. Epub 2014 Apr 16. PMID 24740804
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Lung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; ESC Committee for Practice Guidelines (CPG); Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS). Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2012 Oct;42(4):S1-44. doi: 10.1093/ejcts/ezs455. Epub 2012 Aug 25. No abstract available. PMID 22922698